CLINICAL TRIAL: NCT00061659
Title: A Phase II Randomized Study Evaluating the Safety and Efficacy of ABT-510 in Subjects With Locally Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Study Evaluating the Safety and Efficacy of ABT-510 in Subjects With Locally Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M02-534
Record Dates: First submitted 2003-06-02; First posted 2003-06-04 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Sarcoma, Soft Tissue
Keywords: high grade locally advanced/metastatic soft tissue sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-510 - Thrombospondin-1 mimetic

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of ABT-510 in subjects with locally advanced or metastatic soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for study participation if all of the following criteria are met:

* The subject is at least 18 years of age.
* The subject has histologically confirmed high grade locally advanced or metastatic soft tissue sarcoma (excluding Ewings sarcoma and chondrosarcoma) not amenable to surgery, radiotherapy or combined modality therapy with curative intent.
* The subject must have at least one lesion with measurable disease by RECIST criteria using CT or MRI.
* The subject has received no more than two cytotoxic treatment regimens, not including adjuvant therapy for sarcoma.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
* The subject is able to self-administer or has a caregiver who can reliably administer subcutaneous injections.
* The subject must have adequate bone marrow, renal and hepatic function as follows:

  * Bone marrow: White blood cell count (WBC) greater than or equal to 3,000/mm3; Platelets; greater than or equal to 100,000/mm3; Hemoglobin greater than or equal to 9.0 g/dL;
  * Renal function: Serum creatinine less than or equal to 2.0 mg/dL;
  * Hepatic function: Bilirubin less than or equal to 1.5 mg/dL; AST and ALT less than or equal to 1.5 X the upper normal limit (ULN) unless liver metastases are present, then AST and ALT less than or equal to 5.0 x ULN.
* The subject must not be pregnant or lactating and all subjects (male and female) must use a contraceptive method deemed acceptable by the investigator while in the study and for up to two months following completion of therapy.
* The subject has voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent prior to any study specific procedures.

Exclusion Criteria

A subject will be ineligible for study participation if any of the following criteria are met:

* The subject has a history of or currently exhibits Central Nervous System (CNS) metastasis. Brain MRI within 28 days of enrollment is required to confirm absence of CNS metastases
* The subjects is receiving therapeutic anticoagulation therapy. Low dose anticoagulation (e.g. low dose Coumadin) for catheter prophylaxis will be permitted; PT/PTT must be within normal limits.
* The subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g. hemoptysis). The subject has a recent history (within 4 weeks of Study Day 1) or currently exhibits other clinically significant signs of bleeding.
* The subject has received any therapy for sarcoma including chemotherapy, radiotherapy or any investigational therapy.
* The subject exhibits evidence of clinically significant uncontrolled condition(s) and/or is considered by the investigator to be unable to tolerate the proposed treatment or procedures.
* The subject has history of other previous malignancies within five years, with the exception of:Adequately treated in situ carcinoma of the cervix uteri; Basal or squamous cell carcinoma of the skin.
* The subject's life expectancy is less than 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-05; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival | One year

SECONDARY OUTCOMES:
Response rate | One year
Overall survival | One year
Performance status | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rod Humerickhouse, MD, Study Director — Abbott
Locations (5):
- United States (5):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Center for Sarcoma and Bone Oncology Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cancer Therapy and Research Center, San Antonio, Texas